CLINICAL TRIAL: NCT06827119
Title: Investigation of the Relationship Between Lower Limb Prosthesis Usage Skills and Adaptation Level with Functional Mobility and Activities of Daily Living
Brief Title: Relationship Between Prosthesis Adaptation and Functional Mobility
Status: Completed | Type: Observational
Sponsor: Ankara City Hospital Bilkent (Other)
Responsible Party: Sponsor
Other Study IDs: E2-23-4575
Record Dates: First submitted 2025-02-03; First posted 2025-02-14 (Actual); Last update posted 2025-02-14 (Actual); Status verified 2025-02

CONDITIONS: Amputees / Rehabilitation
Keywords: Earthquake; Amputees; Gait Analysis; Balance

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Cases: Earthquake survivor amputees

SUMMARY:
This study investigates the relationships between locomotor skills, timed performance, gait parameters, balance, fear of falling, and prosthesis satisfaction in individuals who underwent amputation due to an earthquake. Conducted at Ankara Bilkent City Hospital, it included participants aged 18 years and older who were in the prosthetic rehabilitation phase and classified at or above the K1 functional level.

DETAILED DESCRIPTION:
Lower limb amputation significantly affects an individual's mobility, balance, and overall quality of life. The impact is even more pronounced in individuals who have undergone amputation due to traumatic events such as earthquakes. Understanding the factors influencing locomotor performance, balance, and prosthesis satisfaction in this specific population is crucial for optimizing rehabilitation strategies and improving functional outcomes.

This study was conducted at Ankara Bilkent City Hospital and included participants aged 18 years and older, who were in the prosthetic rehabilitation phase and classified at or above the K1 functional level. Participants underwent a series of assessments related to gait, balance, locomotor skills, timed performance, and prosthesis satisfaction. Data were analyzed using correlation analyses, taking into account normality distribution.

The study contributes to the existing literature by highlighting the importance of comprehensive rehabilitation programs that address both physical and psychological aspects of prosthesis adaptation. Future research should focus on larger sample sizes, longer follow-up periods, and the influence of psychosocial factors and rehabilitation approaches on prosthesis satisfaction and functional outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Being over 18 years old
* Having a lower extremity amputation
* Being in the prosthetic period
* Being at K1 functional level or above
* Agreeing to participate in the study voluntarily

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: People admitted to Ankara Bilkent City Hospital
Sampling Method: Non-Probability Sample
Enrollment: 18 (Actual)
Dates: Start 2023-07-19 (Actual); Primary Completion 2024-07-19 (Actual); Study Completion 2024-07-19 (Actual)

PRIMARY OUTCOMES:
K level clasification | Assessed at a single study visit during the 12-month study period.
  The K-level classification was developed by the Centers for Medicare and Medicaid Services (CMS) to determine the current and potential functional mobility levels of prosthetic users. This system rates individuals from K0 (no ability or potential for ambulation with a prosthesis) to K4 (able to use a prosthesis in high-level activities), and it is used as a standardized assessment tool in the prosthetic prescription and reimbursement processes.

OTHER OUTCOMES:
Body Mass Index (BMI): | Assessed at a single study visit during the 12-month study period.
  A calculation based on weight and height to categorize individuals as underweight, normal weight, overweight, or obese.
Joint Range of Motion (ROM): | Assessed at a single study visit during the 12-month study period.
  Measures the movement capability of a joint in degrees, assessing flexibility and any restrictions in motion.
Manuel muscle test | Assessed at a single study visit during the 12-month study period.
  The manual muscle test (MMT) is a clinical method used to evaluate the strength of specific muscles or muscle groups. It involves applying resistance to a muscle's voluntary contraction and grading its performance based on strength and endurance.Typically scored on a 0-5 scale.
Timed Up and Go Test (TUG) | Assessed at a single study visit during the 12-month study period.
  Evaluates functional mobility by measuring the time taken to stand up, walk 3 meters, turn, and return to the chair.
10-Meter Walk Test (10MWT) | Assessed at a single study visit during the 12-month study period.
  Assesses walking speed by timing a person walking a 10-meter distance.
2-Minute Walk Test (2MWT) | Assessed at a single study visit during the 12-month study period.
  Measures endurance by evaluating the distance walked in two minutes.
Houghton Scale | Assessed at a single study visit during the 12-month study period.
  Evaluates prosthesis use and mobility in individuals with lower limb amputations.
Locomotor Capabilities Index (LCI) | Assessed at a single study visit during the 12-month study period.
  A questionnaire that assesses functional mobility, especially in individuals with prosthetic limbs.
Berg Balance Scale (BBS) | Assessed at a single study visit during the 12-month study period.
  A 14-item scale used to measure balance and risk of falling in individuals.
Fear of Falling Visual Analog Scale | Assessed at a single study visit during the 12-month study period.
  A subjective measure of the fear of falling, rated on a 0-10 scale.
Quebec User Evaluation of Satisfaction with Assistive Technology 2.0 (QUEST 2.0) | Assessed at a single study visit during the 12-month study period.
  A questionnaire evaluating user satisfaction with assistive devices in terms of performance and service quality.
Center of Mass (COM) Assessment | Assessed at a single study visit during the 12-month study period.
  Analyzes body balance and stability by tracking COM movements on a specialized platform.
Cadence Measurement with Treadmill-Based Gait Analysis | Assessed at a single study visit during the 12-month study period.
  Uses treadmill equipment to assess cadence (number of steps per minute)
Double Support Percentage Measurement with Treadmill-Based Gait Analysis | Assessed at a single study visit during the 12-month study period.
  Uses treadmill equipment to assess the percentage of time both feet are in contact with the ground during walking
Stride Length Measurement with Treadmill-Based Gait Analysis | Assessed at a single study visit during the 12-month study period.
  Uses treadmill equipment to assess the length of a single stride during walking.
Step Width Measurement with Treadmill-Based Gait Analysis | Assessed at a single study visit during the 12-month study period.
  Uses treadmill equipment to assess the distance between the heels of the feet during walking

CONTACTS AND LOCATIONS:
Locations (1):
- Ankara Bilkent City Hospital, Ankara, Çankaya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Batten HR, McPhail SM, Mandrusiak AM, Varghese PN, Kuys SS. Gait speed as an indicator of prosthetic walking potential following lower limb amputation. Prosthet Orthot Int. 2019 Apr;43(2):196-203. doi: 10.1177/0309364618792723. Epub 2018 Aug 16. PMID 30112982
- [Background] Wong CK, Chen CC, Benoy SA, Rahal RT, Blackwell WM. Role of balance ability and confidence in prosthetic use for mobility of people with lower-limb loss. J Rehabil Res Dev. 2014;51(9):1353-64. doi: 10.1682/JRRD.2013.11.0235. PMID 25785790
- [Background] Zhang X, Liu Z, Qiu G. Measuring Balance Abilities of Transtibial Amputees Using Multiattribute Utility Theory. Biomed Res Int. 2021 Dec 21;2021:8340367. doi: 10.1155/2021/8340367. eCollection 2021. PMID 34970628
- [Background] Abou L, de Freitas GR, Palandi J, Ilha J. Clinical Instruments for Measuring Unsupported Sitting Balance in Subjects with Spinal Cord Injury: A Systematic Review. Top Spinal Cord Inj Rehabil. 2018 Spring;24(2):177-193. doi: 10.1310/sci17-00027. Epub 2018 Feb 12. PMID 29706762
- [Background] Quinzanos-Fresnedo J, Fratini-Escobar PC, Almaguer-Benavides KM, Aguirre-Guemez AV, Barrera-Ortiz A, Perez-Zavala R, Villa-Romero AR. Prognostic validity of a clinical trunk control test for independence and walking in individuals with spinal cord injury. J Spinal Cord Med. 2020 May;43(3):331-338. doi: 10.1080/10790268.2018.1518124. Epub 2018 Sep 12. PMID 30207875
- [Background] Arifin N, Abu Osman NA, Ali S, Gholizadeh H, Abas WA. Postural stability characteristics of transtibial amputees wearing different prosthetic foot types when standing on various support surfaces. ScientificWorldJournal. 2014;2014:856279. doi: 10.1155/2014/856279. Epub 2014 Jun 5. PMID 25003155
- [Background] Wirz M, Muller R, Bastiaenen C. Falls in persons with spinal cord injury: validity and reliability of the Berg Balance Scale. Neurorehabil Neural Repair. 2010 Jan;24(1):70-7. doi: 10.1177/1545968309341059. Epub 2009 Aug 12. PMID 19675123
- [Background] Sahin F, Yilmaz F, Ozmaden A, Kotevolu N, Sahin T, Kuran B. Reliability and validity of the Turkish version of the Berg Balance Scale. J Geriatr Phys Ther. 2008;31(1):32-7. doi: 10.1519/00139143-200831010-00006. PMID 18489806
- [Background] van Ooijen MW, Heeren A, Smulders K, Geurts AC, Janssen TW, Beek PJ, Weerdesteyn V, Roerdink M. Improved gait adjustments after gait adaptability training are associated with reduced attentional demands in persons with stroke. Exp Brain Res. 2015 Mar;233(3):1007-18. doi: 10.1007/s00221-014-4175-7. Epub 2014 Dec 24. PMID 25537466
- [Background] Deathe AB, Wolfe DL, Devlin M, Hebert JS, Miller WC, Pallaveshi L. Selection of outcome measures in lower extremity amputation rehabilitation: ICF activities. Disabil Rehabil. 2009;31(18):1455-73. doi: 10.1080/09638280802639491. PMID 19479574
- [Background] Jackson AB, Carnel CT, Ditunno JF, Read MS, Boninger ML, Schmeler MR, Williams SR, Donovan WH; Gait and Ambulation Subcommittee. Outcome measures for gait and ambulation in the spinal cord injury population. J Spinal Cord Med. 2008;31(5):487-99. doi: 10.1080/10790268.2008.11753644. PMID 19086706
- [Background] Bolliger M, Blight AR, Field-Fote EC, Musselman K, Rossignol S, Barthelemy D, Bouyer L, Popovic MR, Schwab JM, Boninger ML, Tansey KE, Scivoletto G, Kleitman N, Jones LAT, Gagnon DH, Nadeau S, Haupt D, Awai L, Easthope CS, Zorner B, Rupp R, Lammertse D, Curt A, Steeves J. Lower extremity outcome measures: considerations for clinical trials in spinal cord injury. Spinal Cord. 2018 Jul;56(7):628-642. doi: 10.1038/s41393-018-0097-8. Epub 2018 Apr 27. PMID 29700477
- [Background] Martinez-Martin E, Cazorla M. Rehabilitation Technology: Assistance from Hospital to Home. Comput Intell Neurosci. 2019 Jun 2;2019:1431509. doi: 10.1155/2019/1431509. eCollection 2019. PMID 31281333
- [Background] Franchignoni F, Orlandini D, Ferriero G, Moscato TA. Reliability, validity, and responsiveness of the locomotor capabilities index in adults with lower-limb amputation undergoing prosthetic training. Arch Phys Med Rehabil. 2004 May;85(5):743-8. doi: 10.1016/j.apmr.2003.06.010. PMID 15129398
- [Background] Hordacre B, Birks V, Quinn S, Barr C, Patritti BL, Crotty M. Physiotherapy rehabilitation for individuals with lower limb amputation: a 15-year clinical series. Physiother Res Int. 2013 Jun;18(2):70-80. doi: 10.1002/pri.1529. Epub 2012 Jun 6. PMID 22674875
- [Background] Hamamura S, Chin T, Kuroda R, Akisue T, Iguchi T, Kohno H, Kitagawa A, Tsumura N, Kurosaka M. Factors affecting prosthetic rehabilitation outcomes in amputees of age 60 years and over. J Int Med Res. 2009 Nov-Dec;37(6):1921-7. doi: 10.1177/147323000903700630. PMID 20146892
- [Background] Fajardo-Martos I, Roda O, Zambudio-Periago R, Bueno-Cavanillas A, Hita-Contreras F, Sanchez-Montesinos I. Predicting successful prosthetic rehabilitation in major lower-limb amputation patients: a 15-year retrospective cohort study. Braz J Phys Ther. 2018 May-Jun;22(3):205-214. doi: 10.1016/j.bjpt.2017.08.002. Epub 2017 Nov 7. PMID 29157737
- [Background] Hussain E, Kalaycioglu S, Milliner CWD, Cakir Z. Preconditioning the 2023 Kahramanmaras (Turkiye) earthquake disaster. Nat Rev Earth Environ. 2023;4(5):287-289. doi: 10.1038/s43017-023-00411-2. Epub 2023 Apr 24. PMID 37168360
- [Background] McDonald CL, Westcott-McCoy S, Weaver MR, Haagsma J, Kartin D. Global prevalence of traumatic non-fatal limb amputation. Prosthet Orthot Int. 2021 Apr 1;45(2):105-114. doi: 10.1177/0309364620972258. PMID 33274665